CLINICAL TRIAL: NCT00608296
Title: Functional and Neurochemical Brain Changes Following Successful Treatment of Early Course Bipolar Depression
Brief Title: Functional and Neurochemical Brain Changes Bipolar Depression
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Caleb M. Adler, Associate Professor, University of Cincinnati
Other Study IDs: BITREC - Project II
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Study subjects on lithium
- 2: study subjects on quetiapine

SUMMARY:
The purpose of the research is to study brain structure, function and chemistry of patients with bipolar disorder who are receiving quetiapine or lithium, in order to better understand who benefits from treatment and why they respond to medications.

ELIGIBILITY:
Inclusion Criteria - Depressed bipolar patients (N=100; 15-20 patients/year):

1. Patients will meet DSM-IV criteria for type I bipolar disorder, depressed, as determined by structured interview and best-estimate diagnostic procedures.138
2. Patient has experienced a maximum of three documented affective episodes.
3. Patient has been off medications for one week prior to study enrollment.
4. Patient has a Hamilton Depression Rating Scale (HDRS) total score ≥20
5. Patient is between the ages of 12 and 35 years.

Exclusion criteria: All subjects will be excluded from participation for the following reasons:

1. Any chemical use disorder within 3 months.
2. Any history of significant suicidality that would place the patient at risk to participate in this protocol.
3. Current score ≥3 on item 3 of the HDRS-17 (Suicide Item)
4. Any medical or neurological disorder that could influence fMRI results.
5. A history of mental retardation or an estimated IQ total score <85.
6. An MRI scan is contraindicated in the subject for any reason.
7. The patient lives >100 miles from the University of Cincinnati or cannot attend follow-up visits.
8. Meets DSM-IV criteria for a bipolar mixed episode

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: You are being asked to take part in this research study because you have been diagnosed with bipolar disorder and are currently experiencing a depressive episode. Bipolar disorder is an illness characterized by recurrent mood swings including mania, (periods of elation, excessive excitement, irritability, high energy, racing thoughts, poor sleep, poor judgment, reckless behavior) and clinical depression (periods of depressed mood, loss of interest in activities and disruption of sleep, appetite and energy). To participate in this study you must be at least 12 years old, and no older than 35.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caleb M Adler, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States